CLINICAL TRIAL: NCT02771002
Title: Evaluation of the Clinical Assessment of Peripheral Perfusion by Capillary Refill Time and Peripheral Perfusion Index
Brief Title: Assessment of Peripheral Perfusion in the Critically Ill Patient
Acronym: CRTPPI
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: CRTPPI 04/16
Record Dates: First submitted 2016-05-02; First posted 2016-05-12 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Peripheral Perfusion
Keywords: critically ill patients; septic shock; peripheral perfusion index; capillary refill time; mottling score; microcirculation
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood samples for detecting lactate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- septic shock patients: measurements of peripheral perfusion including capillary refill time, mottling score, temperature gradient and peripheral perfusion index hourly until normalisation of lactate sonographic assesment of perfusion of solid organs once within 24h after admission
  Interventions: Device: Peripheral Perfusion index by Carescape Patientenmonitor
- patients rewarming after cardiac surgery: measurements of peripheral perfusion including capillary refill time, mottling score, temperature gradient and peripheral perfusion index hourly until extubation
  Interventions: Device: Peripheral Perfusion index by Carescape Patientenmonitor
- healthy volunteers: measurements of peripheral perfusion including capillary refill time and peripheral perfusion index in ambient temperature and after cooling of extremity
  Interventions: Device: Peripheral Perfusion index by Carescape Patientenmonitor

INTERVENTIONS:
Device: Peripheral Perfusion index by Carescape Patientenmonitor — Peripheral Perfusion index measured with pulse-oximetry by Carescape Patientenmonitor

SUMMARY:
The purpose of this study is to evaluate PPI as a surrogate for clinical signs of peripheral perfusion in patients in septic shock and after cardiac surgery.

DETAILED DESCRIPTION:
The aim of this study is to validate PPI as a continuous, objective measurement of peripheral perfusion indicated by clinical sings of tissue perfusion in patients with septic shock. Furthermore, PPI shall be compared to the perfusion of solid organs evaluated by ultrasound of liver, kidney and gut. In a group of healthy volunteers the investigators will determine normal values in ambient temperature and after cooling of an extremity. Another group of patients after cardiac surgery, where usually a poor tissue perfusion without metabolic failure is present will serve as another "control" population in their post-surgery stabilization period. The values from healthy volunteers and cardiac surgery patients will be compared to those of patients in septic shock.

ELIGIBILITY:
Septic patient:

Inclusion criteria:

* ICU admission with septic shock defined as:
* documented infection (suspected or confirmed) AND
* systemic mean blood pressure <65mmHg requiring any dose of vasopressor despite adequate fluid resuscitation (min. 20ml/kg crystalloids) AND
* lactate >2mmol/l
* Deferred consent by a relative with following informed consent by patient as documented by signatures (Appendix Informed Consent Form)

Exclusion criteria:

* Age <18 or >80 years
* present or suspected myocardial ischemia
* acute pulmonary embolism
* known liver disease - Child-Pugh -Class B or C
* known chronic renal failure
* known peripheral artery disease

Patient after cardiac surgery:

Inclusion criteria:

* ICU admission after coronary artery bypass grafting or valve surgery with cardiopulmonary bypass
* General consent with admission at the University hospital

Exclusion criteria:

* Age <18 or >80 years
* known peripheral artery disease
* no or only low dose of vasopressors (<300µg/h) at ICU admission
* present or suspected myocardial ischemia
* acute pulmonary embolism
* known liver disease - Child-Pugh -Class B or C
* known chronic renal failure

Healthy volunteers:

Inclusion criteria:

- Informed consent as documented by signature (Appendix Informed Consent Form)

Exclusion criteria:

* Age <18 or >80 years
* known peripheral artery disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male septic shock patients with ICU admission Female and male patients after cardiac surgery with ICU admission healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
peripheral perfusion index | measurement at ICU admission and hourly till extubation or normalization of lactate, during the hospitalization without follow-up (maximal up to 72h)
  PPI in healthy controls, septic shock patients and patients rewarming after cardiac surgery

SECONDARY OUTCOMES:
capillary refill time | measurement at ICU admission and hourly till extubation or normalization of lactate, during the hospitalization without follow-up (maximal up to 72h)
  CRT in healthy controls, septic shock patients and patients rewarming after cardiac surgery

OTHER OUTCOMES:
sonographic assesment of solid organ perfusion | within 24h after ICU admission and 24h after first measurement
  solid organ perfusion measured by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No